CLINICAL TRIAL: NCT06586489
Title: The Effects of Virtual Natural Environments in Improving Older Residents' Physical and Psychological Health in Long-term Care Facilities
Brief Title: The Effects of Virtual Natural Environments on Residents' Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202304015
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Psychological Health
Keywords: Virtual Reality; Natural Environments; Older Adults; Randomized Controlled Trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (VR) (Experimental): Participants in this group will engage with immersive virtual reality (VR) natural landscapes.
  Interventions: Behavioral: Virtual Reality Natural Landscape Exposure
- Tablet Screen Group (Tab) (Active Comparator): Participants in this group will view natural landscapes on a tablet screen.
  Interventions: Behavioral: Tablet Screen Natural Landscape Exposure
- Control Group (C) (No Intervention): Participants in this group will continue their usual care routine without additional exposure to virtual or screen-based natural environments.

INTERVENTIONS:
Behavioral: Virtual Reality Natural Landscape Exposure — Participants will view immersive virtual natural landscapes using virtual reality (VR) headsets for 10 minutes, three times a week, over eight weeks. They will choose the natural landscapes they wish to visit and admire, allowing for personalized engagement with the virtual environment.
  Arms: Virtual Reality Group (VR)
Behavioral: Tablet Screen Natural Landscape Exposure — Participants will watch immersive virtual natural landscapes on a tablet screen for 10 minutes, three times a week, over eight weeks. Participants can select the natural landscapes they prefer to view during the sessions, providing a personalized experience.
  Arms: Tablet Screen Group (Tab)

SUMMARY:
This randomized controlled trial aims to explore the impact of virtual natural environments on the mental and physical health of older adults in long-term care facilities. A total of 120 participants will be divided into three groups: a virtual reality (VR) group, a tablet screen-based natural environments group (Tab), and a control group (C) receiving routine care. The intervention involves viewing virtual natural landscapes for 10 minutes, three times a week, over eight weeks. The study will evaluate the effectiveness of these virtual environments in enhancing the quality of life for elderly residents, with data collection occurring at multiple time points. Additionally, qualitative interviews will be conducted with VR group participants to capture their experiences and emotional responses.

DETAILED DESCRIPTION:
This study investigates whether virtual natural environments can improve the mental and physical health of older adults living in long-term care facilities. The trial will involve 120 participants randomly assigned to one of three groups: a virtual reality (VR) group, a tablet screen-based natural environments group (Tab), and a control group (C) receiving routine care. The intervention consists of viewing virtual natural landscapes for 10 minutes, three times a week, over an eight-week period.

The study's primary focus is to assess the impact of these virtual environments on participants' overall well-being and quality of life. Data will be collected at multiple stages throughout the intervention, and statistical analysis will be conducted to determine the effectiveness of the virtual nature sessions. In addition to the quantitative analysis, qualitative interviews will be carried out with participants in the VR group to gather deeper insights into their experiences and the emotional benefits they may derive from the intervention. These interviews will provide valuable context to the quantitative findings, helping to understand the broader implications of using virtual natural environments in long-term care settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Residency in a long-term care institution for more than 1 month
* Clear consciousness

Exclusion Criteria:

* Blindness
* Presence of an infectious disease
* Inability to wear glasses

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Level of Relaxation | Immediately before and immediately after each intervention session
  This study will use the Visual Analogue Scale (VAS) for relaxation.The VAS is a 0-100 mm scale, with 0 mm indicating no relaxation and 100 mm indicating a high level of relaxation.
Temperature | Immediately before and immediately after each intervention session.
  Measurement of body temperature to monitor physiological changes. Unit of Measure: Degrees Celsius (°C)
Heart Rate | Immediately before and immediately after each intervention session.
  Measurement of heart rate to monitor physiological changes. Unit of Measure: Beats per minute (bpm)
Respiration Rate | Immediately before and immediately after each intervention session.
  Measurement of respiration rate to monitor physiological changes. Unit of Measure: Breaths per minute
Blood Pressure | Immediately before and immediately after each intervention session.
  Measurement of blood pressure to monitor physiological changes. Unit of Measure: Millimeters of mercury (mmHg)
Well-being | Baseline (pre-intervention), mid-intervention (week 4), end of intervention (week 8), and follow-up at one month post-intervention (week 12)
  This study will use the 10-item version of the Chinese Happiness Inventory (CHI), adapted from the Oxford Happiness Inventory. The scale has 10 items scored on a 4-point Likert scale, ranging from 0 (minimum) to 3 (maximum), with a total score between 0 and 30. Higher scores indicate greater happiness among elderly residents.
Heart Rate Variability (HRV) | Immediately before and immediately after each intervention session
  HRV refers to the variation in the intervals between heartbeats (RR interval) and is influenced by both the sympathetic and parasympathetic nervous systems. This study will use the VIPcare Plus Smart Band to collect HRV data, including low frequency (LF) and high frequency (HF) power values, as well as the LF/HF ratio, to assess autonomic nervous system balance
Emotion | Baseline (pre-intervention), mid-intervention (week 4), end of intervention (week 8), and follow-up at one month post-intervention (week 12)
  This study will use the Positive and Negative Emotion Scale to measure the emotional states of residents. The scale has 12 items divided into two subscales: the first 6 items assess positive emotions, and the last 6 items assess negative emotions. It is scored on a 5-point Likert scale. The total score for the Positive Emotion Subscale ranges from 6 to 30, where higher scores indicate stronger positive emotions. The Negative Emotion Subscale has the same score range.
Affect | Baseline (pre-intervention), mid-intervention (week 4), end of intervention (week 8), and follow-up at one month post-intervention (week 12)
  The Positive and Negative Affect Schedule (PANAS) will be used to measure emotional states. The scale has 20 items, with 10 items each for positive and negative affect. Higher scores on the Positive Affect Subscale (10-50) indicate higher positive affect, and higher scores on the Negative Affect Subscale (10-50) indicate higher negative affect.
Anxiety | Baseline (pre-intervention), mid-intervention (week 4), end of intervention (week 8), and follow-up at one month post-intervention (week 12)
  The Geriatric Anxiety Inventory (GAI) will be used to assess anxiety levels in elderly residents.The inventory has 20 items, with scores of 0 (no symptoms) or 1 (symptoms present), yielding a total score between 0 and 20. Higher scores indicate higher levels of anxiety.
Perceived Stress | Baseline (pre-intervention), mid-intervention (week 4), end of intervention (week 8), and follow-up at one month post-intervention (week 12)
  The Perceived Stress Scale (PSS-10) will be used to measure the residents perceived stress levels.
Depression | Baseline (pre-intervention), mid-intervention (week 4), end of intervention (week 8), and follow-up at one month post-intervention (week 12)
  The Geriatric Depression Scale-Short Form (GDS-SF) will be used to measure depression levels. The scale consists of 15 items with yes/no responses. The total score ranges from 0 to 15, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Yeu-Hui Chuang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data from this study.